CLINICAL TRIAL: NCT00735527
Title: Intra-Nasal vs. Intra-Venous Lorazepam for Control of Acute Seizures in Children: Prospective Open Labeled Randomized Equivalence Trial
Brief Title: Nasal Versus Venous Lorazepam for Control of Acute Seizures in Children
Acronym: INLOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Ravindra Arya, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INLOR
Record Dates: First submitted 2008-08-12; First posted 2008-08-15 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Status Epilepticus; Seizures
Keywords: seizures; status epilepticus; lorazepam; intra-nasal
MeSH Terms: conditions — Status Epilepticus; Seizures | interventions — Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intra-nasal lorazepam 0.1 mg/kg (max 4 mg)
  Interventions: Drug: Lorazepam
- 2 (Active Comparator): Intra-venous lorazepam 0.1 mg/kg (max 4 mg)
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam — Intra-nasal 0.1 mg/kg (maximum 4 mg) once
  Arms: 1
Drug: Lorazepam — Intra-venous 0.1 mg/kg (maximum 4 mg) once
  Arms: 2

SUMMARY:
Status epilepticus (SE) is a common pediatric emergency which is potentially life-threatening and requires rapid termination. Early and effective treatment is essential to prevent the morbidity and mortality associated with prolonged convulsive SE. Lorazepam is the standard of care for control of SE when administered by intra-venous (IV) route. The investigators intend to compare efficacy and adverse effect profile of intra-nasal vs. intravenous routes of administration of lorazepam. In resource poor settings, sometimes trained personnel or appropriate equipment for intra-venous cannulation is not available. Alternate routes of administration, if shown equivalent to conventional IV route, will be very useful in such settings or for out of hospital management of seizures in children.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting convulsing to the pediatric emergency or developing seizure while in casualty
* Age 6-14 years

Exclusion Criteria:

* Known hypersensitivity to any benzodiazepine
* Child has received any parenteral anti-convulsant within 1 hr prior to enrollment
* Presence of severe cardio-respiratory compromise or cardiac arrhythmias
* Presence of upper respiratory tract infection
* Presence of basal skull fracture causing cerebro-spinal fluid (CSF) rhinorrhea

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Cessation of all clinical seizure activity within 10 min of drug administration | 10 min

SECONDARY OUTCOMES:
Persistent cessation of seizure activity for 1 hr | 1 hr
Patients requiring rescue medication within 1 hr | 1 hr
Time to achieve intra-venous access after arrival in casualty | minutes
Time from drug administration to termination of seizure(s) | minutes
Development of hypotension (fall of >/= 20 mmHg systolic and/ or >/= 10 mmHg diastolic pressure) within 1 hr of drug administration | 1 hr
Development of significant respiratory depression requiring assisted ventilation | 1 hr

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Arya R, Gulati S, Kabra M, Sahu JK, Kalra V. Intranasal versus intravenous lorazepam for control of acute seizures in children: a randomized open-label study. Epilepsia. 2011 Apr;52(4):788-93. doi: 10.1111/j.1528-1167.2010.02949.x. Epub 2011 Jan 28. PMID 21275979